CLINICAL TRIAL: NCT06844981
Title: Moviendo Las Caderas: Effects of Latin Dancing on Sleep Quality in Hispanic Cancer Survivors
Brief Title: Effects of Latin Dancing on Sleep Quality in Hispanic Cancer Survivors
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Evelyn Arana, DrPH, Assistant Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Pro2025000098
Record Dates: First submitted 2025-01-28; First posted 2025-02-25 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Cancer Survivorship; Sleep Disturbances
Keywords: Cancer; Cancer Survivorship; Sleep Disturbances; Hispanic Cancer Survivors; Latin Dancing
MeSH Terms: conditions — Parasomnias; Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care arm (No Intervention): Participants in the usual care arm will receive care as usual and will not participate in the Latin Dancing program.
- Intervention arm (Experimental): Participants in this arm will participate in the virtual Latin Dance group program that meets for 8 weeks, 2x each week, for 75 minute sessions.
  Interventions: Behavioral: Latin Dance

INTERVENTIONS:
Behavioral: Latin Dance — Latin Dance intervention
  Other Names: intervention arm
  Arms: Intervention arm

SUMMARY:
The primary objective is to assess the feasibility, acceptability and explore the impact of a culturally appropriate Latin Dance intervention vs. Usual Care on sleep quality for Hispanic cancer survivors.

Secondary objectives are to examine the preliminary efficacy of a culturally appropriate Latin Dance intervention on secondary cancer- and treatment-related side effects (e.g., Quality of Life, distress, insomnia, fatigue).

DETAILED DESCRIPTION:
In this feasibility Randomized Control Trial (RCT) study, the investigators will assess the feasibility, acceptability, and explore the impact of a Latin dance intervention vs usual care on sleep quality among Hispanic survivors.

Study Aims:

Aim 1: Develop a culturally appropriate Latin dance intervention for Hispanic cancer survivors using a bidirectional community engagement approach. Using iterative qualitative feedback from Hispanic cancer survivors, the investigators will develop a Latin dance intervention for Hispanic cancer survivors.

Aim 2: Assess the feasibility and acceptability of a culturally appropriate Latin Dance intervention for Hispanic cancer survivors.

Aim 3: Provide preliminary evidence of the efficacy potential of a culturally appropriate Latin Dance intervention vs. usual care on subjective and objective sleep quality for Hispanic survivors.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years of age or older
* Self-identify as Hispanic and/or Latino(a)
* Have a confirmed diagnosis of a solid tumor or hematologic malignancy
* Must have completed primary cancer treatment 3+ months prior to enrollment (e.g., chemotherapy, surgery, and/or radiation therapy but may be on hormonal therapy and/or immunotherapy or other long-term therapies)
* Have sleep disturbance (indicated by a response of 3 or more on the MD Anderson Symptom Inventory sleep question by using an 11-point scale anchored by 0 [no sleep disturbance] and 10 [worst possible sleep disturbance]
* Be able to read and understand English and/or Spanish
* Physically Inactive (<150 minutes of vigorous exercise/week within the past 3 months)

Exclusion Criteria:

* Current regular Latin dancing practice within the past year (2-3 times a week over a period of two months that is not interrupted).
* Inability to speak and read English or Spanish proficiently
* Inability to understand informed consent
* Medical conditions that can cause sleep impairment: sleep apnea, restless leg syndrome, shift work
* Regular use of a walker or wheelchair
* Healing or unhealed fractures
* Heart failure
* Life expectancy <12 months
* Unwilling to be randomized to study arms and/or commit to 8 weeks of classes and a follow-up assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the Intervention | 8 weeks
  Feasibility in this study will include recruitment, adherence, and retention rates.
Treatment Perception Questionnaire (Acceptability of Intervention) | Post-intervention (at approximately 8 weeks)
  Acceptability is defined as at least 80% of participants in the Latin Dance group agreeing or strongly agreeing that the intervention was acceptable via the Treatment Perceptions Questionnaire (TPQ). The TPQ consists of 10 statements about treatment satisfaction on a Likert-type scale from 0 (strongly disagree) to 4 (strongly agree). Average scores ≥ 3 indicated acceptable satisfaction.
Pittsburgh Sleep Quality Index | Baseline and post-intervention (approximately 8 weeks)
  Changes in sleep quality will be assessed pre and post-intervention with the Pittsburgh Sleep Quality Index (PSQI). The PSQI measures sleep quality with a total score ranging from 0-21 with higher scores indicating worse sleep quality.

SECONDARY OUTCOMES:
Functional Outcomes for Cancer Therapy - General | Baseline and post-intervention (approximately 8 weeks)
  Quality of Life will be assessed via the Functional Outcomes for Cancer Therapy - General (FACT-G). This measure consists of 27 items designed to measure four domains of quality of life in cancer patients: physical, social, emotional, and functional well-being. Coefficients of reliability and validity are uniformly high. The physical, social, and functional domain scores range from 0-28 with higher scores indicating better quality of life. The emotional domain score ranges from 0 - 24 with higher scores indicating better quality of life. The FACT-G total score ranges from 0 - 108, with higher scores indicating better quality of life.
Functional Assessment of Chronic Illness - Fatigue | Baseline and post-intervention (approximately 8 weeks)
  Fatigue will be assessed with the Functional Assessment of Chronic Illness - Fatigue (FACIT-F) Scale. Higher scores indicate less fatigue (score range=0-52).
Patient Health Questionnaire - 2 (PHQ-2) | Baseline and post-intervention (approximately 8 weeks)
  The PHQ-2 is a two-item screening questionnaire for depression that asks about the frequency of a depressed mood and loss of interest or pleasure in the last two weeks. Each of the two questions is scored from 0 to 3, based on frequency. The two scores are added together for a total score ranging from 0 to 6. A total score of 3 or higher indicates a positive screen for depression.
Generalized Anxiety Disorder - 7 (GAD-7) | Baseline and post-intervention (approximately 8 weeks)
  The GAD-7 is used for screening and measuring the severity of generalized anxiety disorder (GAD). The total score indicates the severity of anxiety, from minimal (0-4) to severe (15 and above)
Insomnia Severity Index | Baseline and post-intervention (approximately 8 weeks)
  Insomnia will be assessed with the Insomnia Severity Index (ISI). A 5-point Likert scale of 7 questions is used to rate each item (e.g., 0 = no problem; 4 = very severe problem), yielding a total score ranging from 0 to 28 with higher scores indicating higher severity of insomnia.
Objective Symptoms of Insomnia- Sleep Duration Via Actigraphy | 2 weeks (worn for 1 week at Baseline and 1 week at post-intervention)
  Actigraphy will measure the number of minutes of actual sleep.
Objective Symptoms of Insomnia- Wake After Sleep Onset Via Actigraphy | 2 weeks (worn for 1 week at Baseline and 1 week at post-intervention)
  Actigraphy will measure total minutes of wake time after sleep onset.
Objective Symptoms of Insomnia- Sleep Efficiency via Actigraphy | 2 weeks (worn for 1 week at Baseline and 1 week at post-intervention)
  Actigraphy will measure the percent of time actually slept compared to intended time sleeping.
Objective Symptoms of Insomnia- Sleep Latency Via Actigraphy | 2 weeks (worn for 1 week at Baseline and 1 week at post-intervention)
  Actigraphy will measure the minutes it takes for the participant to fall asleep.
Charleson Comorbidity Index | Baseline and post-intervention (approximately 8 weeks)
  The Charleson Comorbidity Index consists of 19 items, each with an assigned weight from 1 to 6 according to the relative risk of dying within a year. In general, the absence of comorbidity is considered: 0-1 points; low comorbidity: 2 points; and high comorbidity: ≥3 points.
Physical Activity Daily Diaries | Physical activity daily diaries will be completed beginning 1 week pre-intervention, completed throughout the 8-week intervention, and 1-week post-intervention.
  The physical activity daily diary is designed to gather information about participants' daily physical activity patterns.
Sleep Daily Diaries | Sleep daily diaries will be completed beginning 1 week pre-intervention, completed throughout the 8-week intervention, and 1-week post-intervention.
  The sleep diary is designed to gather information about participants' daily sleep patterns.
Self-Efficacy for Exercise (SEE) Scale | Baseline and post-intervention (approximately 8 weeks)
  The Self-Efficacy for Exercise (SEE) scale is a questionnaire designed to measure an individual's confidence in their ability to exercise regularly. Participants rate their confidence on a scale, often from 0 (not at all confident) to 10 (very confident).
Short Acculturation Scale for Hispanics (SASH) | Baseline
  The Short Acculturation Scale for Hispanics is a 12-item questionnaire developed to measure the degree of acculturation experienced by Hispanics in the United States. Scores range from 1 to 5, where higher scores indicate a greater level of acculturation to mainstream U.S. culture.
Discrimination in Medical Settings Scale | Baseline and post-intervention (approximately 8 weeks)
  The Discrimination in Medical Settings (DMS) scale is a 7-item questionnaire that measures patient-reported experiences of mistreatment in healthcare settings. It uses a 5-point Likert scale for each item, asking patients how often they have experienced specific scenarios, such as being treated with less courtesy or feeling a doctor is not listening to them. Higher scores on the scale indicate more frequent experiences of discrimination, and it is used to study disparities in healthcare.
Brief Pain Inventory (BPI) | Baseline and post-intervention (approximately 8 weeks)
  The Brief Pain Inventory (BPI) is a 9-item self-report tool that measures pain severity and how pain interferes with daily activities on a 0-10 scale, with higher scores indicating greater pain. It shows excellent reliability, with Cronbach's alpha typically between 0.80 and 0.95.
Leisure Time Exercise Questionnaire of Godin and Shephard | Baseline and post-intervention (approximately 8 weeks)
  The Leisure-Time Exercise Questionnaire (LTEQ) by Godin and Shephard is a brief self-report measure that asks about the frequency of mild, moderate, and strenuous exercise during a typical week. Responses are converted into a weekly leisure activity score by weighting each intensity level. The LTEQ demonstrates good reliability, with Cronbach's alpha values around 0.80 and strong test-retest stability.

CONTACTS AND LOCATIONS:
Overall Officials: Evelyn Arana, DrPH, Principal Investigator — Rutgers Cancer Institute
Locations (1):
- Rutgers Cancer Institute, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No